CLINICAL TRIAL: NCT01374425
Title: MAVERICC (Marker Evaluation for Avastin Research in CRC): A Randomized Phase II Study of Bevacizumab+mFOLFOX6 Vs. Bevacizumab+FOLFIRI With Biomarker Stratification in Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: Study of Bevacizumab + mFOLFOX6 Versus Bevacizumab + FOLFIRI With Biomarker Stratification in Participants With Previously Untreated Metastatic Colorectal Cancer (mCRC)
Acronym: MAVERICC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25710; 2011-004755-39 (EudraCT Number)
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Bevacizumab; Irinotecan; Leucovorin; Oxaliplatin; Capecitabine

ARMS (2):
- Bevacizumab + mFOLFOX6 (Experimental): Participants will receive bevacizumab plus mFOLFOX6 by intravenous (IV) infusion on Day 1 of each 2-week cycle until disease progression or unacceptable toxicity. Participants may be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin, with bevacizumab continued in 3-week cycles.
  Interventions: Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Capecitabine
- Bevacizumab + FOLFIRI (Experimental): Participants will receive bevacizumab plus FOLFIRI by IV infusion on Day 1 of each 2-week cycle until disease progression or unacceptable toxicity. Participants may be transitioned to oral capecitabine in the event of unacceptable toxicity to irinotecan, with bevacizumab continued in 3-week cycles.
  Interventions: Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Irinotecan; Drug: Leucovorin; Drug: Capecitabine

INTERVENTIONS:
Drug: 5-Fluorouracil — 5-Fluorouracil 400 milligrams per meter-squared (mg/m^2) by IV bolus and subsequent 2400 mg/m^2 by IV infusion over 46 hours will be administered every 2 weeks until disease progression or unacceptable toxicity.
Drug: Bevacizumab — Bevacizumab 5 milligrams per kilogram (mg/kg) of body weight via IV infusion will be administered every 2 weeks until disease progression or unacceptable toxicity. If participants are discontinued from oxaliplatin or irinotecan due to unacceptable toxicity, bevacizumab may be given in 3-week cycles with capecitabine.
  Other Names: Avastin
Drug: Irinotecan — Irinotecan 180 mg/m^2 via IV infusion over 2 hours will be administered every 2 weeks until disease progression or unacceptable toxicity.
  Arms: Bevacizumab + FOLFIRI
Drug: Leucovorin — Leucovorin 400 mg/m^2 or dose deemed appropriate by Investigator via IV infusion over 2 hours will be administered every 2 weeks until disease progression or unacceptable toxicity.
Drug: Oxaliplatin — Oxaliplatin 85 mg/m^2 via IV infusion over 2 hours will be administered every 2 weeks until disease progression or unacceptable toxicity.
  Arms: Bevacizumab + mFOLFOX6
Drug: Capecitabine — Capecitabine 850 or 1000 mg/m^2 may be offered in the event of unacceptable toxicity to oxaliplatin or irinotecan, to be given orally twice a day on Days 1 to 14 in 3-week cycles.

SUMMARY:
This will be a randomized, open-label, multicenter, Phase II study with primary objectives to assess whether expression of select chemotherapy markers is associated with progression-free survival (PFS) in participants treated with bevacizumab plus leucovorin, 5-fluorouracil, and oxaliplatin (mFOLFOX6) or bevacizumab plus leucovorin, 5-fluorouracil, and irinotecan (FOLFIRI). The study population will consist of participants with first-line mCRC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed colorectal cancer (CRC) with at least one measurable metastatic lesion by RECIST Version 1.1
* Archival tumor tissue sample must be requested and available prior to study entry. If no archival tumor tissue sample is available, a fresh biopsy tissue sample must be obtained but should be discussed first with the medical monitor. A copy of the local pathology report must be submitted along with the specimens.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participants with treated brain metastases are eligible for study participation. Participants may not receive ongoing treatment with steroids at Screening. Anticonvulsants (at stable dose) are allowed. Treatment for brain metastases may be whole-brain radiotherapy, radiosurgery, neurosurgery, or a combination as deemed appropriate by the treating physician. Radiotherapy and stereotactic radiosurgery must be completed at least 28 days prior to randomization.
* Female participants should not be pregnant or breastfeeding. Female participants with childbearing potential should agree to use effective, non-hormonal means of contraception during the study and for a period of at least 6 months following the last administration of study drugs. Female participants with an intact uterus (unless amenorrheic for the last 24 months) must have a negative serum pregnancy test within 7 days prior to randomization into the study.
* Male participants must agree to use effective contraception during the study and for a period of at least 6 months following the last administration of study drugs, even if they have been surgically sterilized.

Exclusion Criteria:

* Any prior systemic treatment for mCRC
* Adjuvant chemotherapy for CRC completed <12 months
* Evidence of Gilbert's syndrome or of homozygosity for the UGT1A1*28 allele
* Known positivity for human immunodeficiency virus (HIV)
* Malignancies other than mCRC within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, and ductal carcinoma in situ treated surgically with curative intent
* Radiotherapy to any site for any reason within 28 days prior to randomization, except for palliative radiotherapy to bone lesions within 14 days prior to randomization
* Clinically detectable third-space fluid collections that cannot be controlled by drainage or other procedures prior to study entry
* Treatment with any other investigational agent, or participation in another investigational drug trial within 28 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2011-08; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Langer, M.D., Study Director — Genentech, Inc.
Locations (76):
- United States (62):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Bellflower, California
  - Duarte, California
  - Fountain Valley, California
  - Fresno, California
  - Hayward, California
  - Los Angeles, California
  - Oakland, California
  - Pleasant Hill, California
  - Roseville, California
  - Sacramento, California
  - San Francisco, California
  - San Jose, California
  - Santa Clara, California
  - South San Francisco, California
  - Vallejo, California
  - Walnut Creek, California
  - Denver, Colorado
  - Stamford, Connecticut
  - Trumbull, Connecticut
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Port Saint Lucie, Florida
  - Boise, Idaho
  - Joliet, Illinois
  - Maywood, Illinois
  - Peoria, Illinois
  - Goshen, Indiana
  - Indianapolis, Indiana
  - Terre Haute, Indiana
  - Fairway, Kansas
  - Elizabethtown, Kentucky
  - Scarborough, Maine
  - Burlington, Massachusetts
  - Billings, Montana
  - Lincoln, Nebraska
  - Cherry Hill, New Jersey
  - Manasquan, New Jersey
  - Albuquerque, New Mexico
  - Farmington, New Mexico
  - Las Cruces, New Mexico
  - Santa Fe, New Mexico
  - Rochester, New York
  - Durham, North Carolina
  - Greensboro, North Carolina
  - High Point, North Carolina
  - Washington, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Dunmore, Pennsylvania
  - Media, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Corpus Christi, Texas
  - Houston, Texas
  - Madison, Wisconsin
  - Wauwatosa, Wisconsin
- Edmonton, Alberta, Canada
- Estonia (2):
  - Tallinn
  - Tartu
- Ireland (3):
  - Cork
  - Dublin
  - Galway
- Oslo, Norway
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Switzerland (4):
  - Aarau
  - Basel
  - Lucerne
  - Zurich

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial included a 21-day Screening period during which participants provided information for demographics, medical history, and cancer/treatment history and completed urinalysis collection.
Groups:
- Bevacizumab + mFOLFOX6: Participants with untreated metastatic colorectal cancer (mCRC) who were candidates for first-line therapy received bevacizumab plus leucovorin, 5-fluorouracil, and oxaliplatin (mFOLFOX6) until disease progression or unacceptable toxicity. Bevacizumab was given as 5 milligrams per kilogram (mg/kg), leucovorin as 400 milligrams per meter-squared (mg/m^2), oxaliplatin as 85 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via intravenous (IV) infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles.
- Bevacizumab + FOLFIRI: Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus leucovorin, 5-fluorouracil, and irinotecan (FOLFIRI) until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles.
Period: Overall Study
Arm/Group | Bevacizumab + mFOLFOX6 | Bevacizumab + FOLFIRI
Started | 188 | 188
Completed | 0 | 0
Not Completed | 188 | 188
Not completed — Radiographic Disease Progression | 86 | 81
Not completed — Clinical Disease Progression | 9 | 6
Not completed — Adverse Event | 29 | 18
Not completed — Death (Progression of Disease) | 1 | 0
Not completed — Death (Adverse Event) | 2 | 4
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Refused Treatment | 10 | 24
Not completed — Protocol Violation | 2 | 3
Not completed — Sponsor Decision | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Other | 41 | 43

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All randomized participants regardless of receiving any study drug.
Groups:
- Bevacizumab + mFOLFOX6: Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles.
- Bevacizumab + FOLFIRI: Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + mFOLFOX6 | Bevacizumab + FOLFIRI | Total
Number analyzed (Participants) | 188 | 188 | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (10.88) | 60.7 (10.66) | 59.9 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 71 | 137
  Male | 122 | 117 | 239

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Tumor assessments were performed according to RECIST Version 1.1. Disease progression was defined as greater than or equal to (≥) 20 percent (%) increase in sum of largest diameters (LD) of target lesions in reference to the smallest sum of LD on study, in addition to an absolute increase ≥5 millimeters (mm). Disease progression was further defined as the last documented progression determined by the Investigator no later than 1 day before initiation of second-line therapy. Death on study included death from any cause occurring no later than 3 months after the last component of study treatment. PFS was defined as the time from randomization to death or disease progression, whichever occurred first. The median duration of PFS was estimated by Kaplan-Meier analysis and expressed in months. The 95% confidence interval (CI) was computed using the method of Brookmeyer and Crowley.
Time Frame: From Baseline until death or disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: Intent-to-treat (ITT) Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX6 | Bevacizumab + FOLFIRI
Number analyzed (Participants) | 188 | 188
months | 10.09 [8.80 to 11.56] | 12.55 [10.48 to 14.29]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 vs Bevacizumab + FOLFIRI; Analysis stratified by high/low excision repair cross-complementing (ERCC)-1 level and region of enrollment; Test type: Superiority or Other; p = 0.0555, Log Rank — P-value (relative to Bevacizumab + mFOLFOX6) based on two-sided stratified log rank test and not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.61 to 1.01] — Hazard ratio (HR) (relative to Bevacizumab + mFOLFOX6) was estimated by Cox regression

2. Primary Outcome: PFS According to RECIST Version 1.1 in Participants With High ERCC-1 Levels
Description: Tumor assessments were performed according to RECIST Version 1.1. Disease progression was defined as ≥20% increase in sum of LD of target lesions in reference to the smallest sum of LD on study, in addition to an absolute increase ≥5 mm. Disease progression was further defined as the last documented progression determined by the Investigator no later than 1 day before initiation of second-line therapy. Death on study included death from any cause occurring no later than 3 months after the last component of study treatment. PFS was defined as the time from randomization to death or disease progression, whichever occurred first. The median duration of PFS was estimated by Kaplan-Meier analysis and expressed in months. The 95% CI was computed using the method of Brookmeyer and Crowley.
Time Frame: From Baseline until death or disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: ITT Population. The "Number of Participants Analyzed" reflects the number of evaluable participants for the outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX6 (ERCC-1 High): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level greater than (>) 1.7 × 10^-3 ERCC-1/B-actin messenger ribonucleic acid (mRNA) at Baseline were included in separate analyses.
- Bevacizumab + FOLFIRI (ERCC-1 High): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level >1.7 × 10^-3 ERCC-1/B-actin mRNA at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 High) | Bevacizumab + FOLFIRI (ERCC-1 High)
Number analyzed (Participants) | 64 | 67
months | 9.92 [8.51 to 12.48] | 11.17 [9.10 to 17.84]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 High) vs Bevacizumab + FOLFIRI (ERCC-1 High); Analysis stratified by region of enrollment; Test type: Superiority or Other; p = 0.3944, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.56 to 1.26] — HR (relative to Bevacizumab + mFOLFOX6) was estimated by Cox regression

3. Primary Outcome: PFS According to RECIST Version 1.1 in Participants With Low ERCC-1 Levels
Description: as for outcome 2
Time Frame: From Baseline until death or disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX6 (ERCC-1 Low): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level less than or equal to (≤) 1.7 × 10^-3 ERCC-1/B-actin mRNA at Baseline were included in separate analyses.
- Bevacizumab + FOLFIRI (ERCC-1 Low): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level ≤1.7 × 10^-3 ERCC-1/B-actin mRNA at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 Low) | Bevacizumab + FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 124 | 120
months | 10.97 [8.54 to 12.29] | 12.68 [10.48 to 14.49]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 Low) vs Bevacizumab + FOLFIRI (ERCC-1 Low); Analysis stratified by region of enrollment; Test type: Superiority or Other; p = 0.0786, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.55 to 1.03] — HR (relative to Bevacizumab + mFOLFOX6) was estimated by Cox regression

4. Primary Outcome: PFS According to RECIST Version 1.1 in Participants With High ERCC-1 Levels Versus Participants With Low ERCC-1 Levels
Description: as for outcome 2
Time Frame: From Baseline until death or disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 or bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Depending on the regimen to which the participant was randomized, bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin or irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level >1.7 × 10^-3 ERCC-1/B-actin mRNA at Baseline were included in separate analyses.
- Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 or bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Depending on the regimen to which the participant was randomized, bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin or irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level ≤1.7 × 10^-3 ERCC-1/B-actin mRNA at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 131 | 244
months | 10.87 [9.10 to 12.68] | 11.56 [9.95 to 12.98]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) vs Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low); Analysis stratified by region of enrollment; Test type: Superiority or Other; p = 0.9576, Log Rank — P-value (relative to ERCC-1 Low subgroup) based on two-sided stratified log rank test and not adjusted for multiple comparisons; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.77 to 1.28] — HR (relative to ERCC-1 Low subgroup) was estimated by Cox regression

5. Primary Outcome: PFS According to RECIST Version 1.1 in Participants With High Vascular Endothelial Growth Factor (VEGF)-A Levels Versus Participants With Low VEGF-A Levels
Description: as for outcome 2
Time Frame: From Baseline until death or disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 or bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Depending on the regimen to which the participant was randomized, bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin or irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with VEGF-A level >5 picograms per milliliter (pg/mL) at Baseline were included in separate analyses.
- Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 or bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Depending on the regimen to which the participant was randomized, bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin or irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with VEGF-A level ≤5 pg/mL at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low)
Number analyzed (Participants) | 185 | 185
months | 10.02 [8.80 to 11.17] | 12.68 [10.9 to 14.26]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) vs Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low); Analysis stratified by high/low ERCC-1 level and region of enrollment; Test type: Superiority or Other; p = 0.1658, Log Rank — P-value (relative to VEGF-A Low subgroup) based on two-sided stratified log rank test and not adjusted for multiple comparisons; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.93 to 1.53] — HR (relative to VEGF-A Low subgroup) was estimated by Cox regression

6. Secondary Outcome: PFS According to RECIST Version 1.1 in Participants With High ERCC-1 and High VEGF-A Levels
Description: as for outcome 2
Time Frame: From Baseline until death or disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX6 (ERCC-1 High, VEGF-A High): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level >1.7 × 10^-3 ERCC-1/B-actin mRNA and VEGF-A level >5 pg/mL at Baseline were included in separate analyses.
- Bevacizumab + FOLFIRI (ERCC-1 High, VEGF-A High): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level >1.7 × 10^-3 ERCC-1/B-actin mRNA and VEGF-A level >5 pg/mL at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 High, VEGF-A High) | Bevacizumab + FOLFIRI (ERCC-1 High, VEGF-A High)
Number analyzed (Participants) | 28 | 31
months | 8.80 [5.91 to 10.02] | 11.17 [8.11 to 18.07]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 High, VEGF-A High) vs Bevacizumab + FOLFIRI (ERCC-1 High, VEGF-A High); Analysis stratified by region of enrollment; Test type: Superiority or Other; p = 0.3019, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.41 to 1.32] — HR (relative to Bevacizumab + mFOLFOX6) was estimated by Cox regression

7. Secondary Outcome: PFS According to RECIST Version 1.1 in Participants With High ERCC-1 and Low VEGF-A Levels
Description: as for outcome 2
Time Frame: From Baseline until death or disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX6 (ERCC-1 High, VEGF-A Low): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level >1.7 × 10^-3 ERCC-1/B-actin mRNA and VEGF-A level ≤5 pg/mL at Baseline were included in separate analyses.
- Bevacizumab + FOLFIRI (ERCC-1 High, VEGF-A Low): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level >1.7 × 10^-3 ERCC-1/B-actin mRNA and VEGF-A level ≤5 pg/mL at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 High, VEGF-A Low) | Bevacizumab + FOLFIRI (ERCC-1 High, VEGF-A Low)
Number analyzed (Participants) | 35 | 35
months | 12.52 [9.43 to 15.64] | 12.68 [8.18 to 20.83]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 High, VEGF-A Low) vs Bevacizumab + FOLFIRI (ERCC-1 High, VEGF-A Low); Analysis stratified by region of enrollment; Test type: Superiority or Other; p = 0.6035, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.48 to 1.53] — HR (relative to Bevacizumab + mFOLFOX6) was estimated by Cox regression

8. Secondary Outcome: PFS According to RECIST Version 1.1 in Participants With Low ERCC-1 and High VEGF-A Levels
Description: as for outcome 2
Time Frame: From Baseline until death or disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX6 (ERCC-1 Low, VEGF-A High): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level ≤1.7 × 10^-3 ERCC-1/B-actin mRNA and VEGF-A level >5 pg/mL at Baseline were included in separate analyses.
- Bevacizumab + FOLFIRI (ERCC-1 Low, VEGF-A High): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level ≤1.7 × 10^-3 ERCC-1/B-actin mRNA and VEGF-A level >5 pg/mL at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 Low, VEGF-A High) | Bevacizumab + FOLFIRI (ERCC-1 Low, VEGF-A High)
Number analyzed (Participants) | 66 | 59
months | 9.76 [8.18 to 12.45] | 11.07 [8.18 to 14.29]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 Low, VEGF-A High) vs Bevacizumab + FOLFIRI (ERCC-1 Low, VEGF-A High); Analysis stratified by region of enrollment; Test type: Superiority or Other; p = 0.4032, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.54 to 1.28] — HR (relative to Bevacizumab + mFOLFOX6) was estimated by Cox regression

9. Secondary Outcome: PFS According to RECIST Version 1.1 in Participants With Low ERCC-1 and Low VEGF-A Levels
Description: as for outcome 2
Time Frame: From Baseline until death or disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX6 (ERCC-1 Low, VEGF-A Low): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level ≤1.7 × 10^-3 ERCC-1/B-actin mRNA and VEGF-A level ≤5 pg/mL at Baseline were included in separate analyses.
- Bevacizumab + FOLFIRI (ERCC-1 Low, VEGF-A Low): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level ≤1.7 × 10^-3 ERCC-1/B-actin mRNA and VEGF-A level ≤5 pg/mL at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 Low, VEGF-A Low) | Bevacizumab + FOLFIRI (ERCC-1 Low, VEGF-A Low)
Number analyzed (Participants) | 55 | 60
months | 11.10 [8.54 to 13.08] | 14.32 [11.56 to 14.98]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 Low, VEGF-A Low) vs Bevacizumab + FOLFIRI (ERCC-1 Low, VEGF-A Low); Analysis stratified by region of enrollment; Test type: Superiority or Other; p = 0.0647, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.41 to 1.03] — HR (relative to Bevacizumab + mFOLFOX6) was estimated by Cox regression

10. Secondary Outcome: Overall Survival (OS)
Description: Death on study included death from any cause occurring no later than 3 months after the last component of study treatment. OS was defined as the time from randomization to death. The median duration of OS was estimated by Kaplan-Meier analysis and expressed in months. The 95% CI was computed using the method of Brookmeyer and Crowley.
Time Frame: From Baseline until death (maximum up to 45 months overall)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX6 | Bevacizumab + FOLFIRI
Number analyzed (Participants) | 188 | 188
months | 23.85 [20.40 to 26.05] | 27.47 [24.64 to 36.73]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 vs Bevacizumab + FOLFIRI; Analysis stratified by high/low ERCC-1 level and region of enrollment; Test type: Superiority or Other; p = 0.0861, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.56 to 1.04] — HR (relative to Bevacizumab + mFOLFOX6) was estimated by Cox regression

11. Secondary Outcome: OS in Participants With High ERCC-1 Levels
Description: as for outcome 10
Time Frame: From Baseline until death (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX6 (ERCC-1 High): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level >1.7 × 10^-3 ERCC-1/B-actin mRNA at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 High) | Bevacizumab + FOLFIRI (ERCC-1 High)
Number analyzed (Participants) | 64 | 67
months | 22.54 [17.02 to 26.05] | 26.51 [19.09 to 36.73]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 High) vs Bevacizumab + FOLFIRI (ERCC-1 High); Analysis stratified by region of enrollment; Test type: Superiority or Other; p = 0.3295, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.51 to 1.26] — HR (relative to Bevacizumab + mFOLFOX6) was estimated by Cox regression

12. Secondary Outcome: OS in Participants With Low ERCC-1 Levels
Description: as for outcome 10
Time Frame: From Baseline until death (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX6 (ERCC-1 Low): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 until disease progression or unacceptable toxicity. Bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with ERCC-1 level ≤1.7 × 10^-3 ERCC-1/B-actin mRNA at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 Low) | Bevacizumab + FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 124 | 120
months | 25.53 [20.40 to 28.75] | 27.93 [24.97 to 38.44]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 Low) vs Bevacizumab + FOLFIRI (ERCC-1 Low); Analysis stratified by region of enrollment; Test type: Superiority or Other; p = 0.1519, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.49 to 1.12] — HR (relative to Bevacizumab + mFOLFOX6) was estimated by Cox regression

13. Secondary Outcome: OS in Participants With High ERCC-1 Levels Versus Participants With Low ERCC-1 Levels
Description: as for outcome 10
Time Frame: From Baseline until death (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 131 | 244
months | 23.23 [19.09 to 26.94] | 27.27 [24.34 to 31.28]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) vs Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low); Analysis stratified by region of enrollment; Test type: Superiority or Other; p = 0.2774, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.87 to 1.62] — HR (relative to ERCC-1 Low subgroup) was estimated by Cox regression

14. Secondary Outcome: Percentage of Participants With Objective Response According to RECIST Version 1.1
Description: Objective response was defined as complete response (CR) or partial response (PR) according to RECIST Version 1.1. CR was defined as disappearance of all target lesions and short-axis reduction to less than (<) 10 mm of any pathological lymph nodes. PR was defined as ≥30% decrease in sum of LD of target lesions in reference to sum of LD at Baseline. Confirmation of response at a consecutive assessment was not required. The percentage of participants with CR or PR was reported. The 95% CI was computed using normal approximation to the binomial distribution.
Time Frame: From Baseline until disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 | Bevacizumab + FOLFIRI
Number analyzed (Participants) | 188 | 188
percentage of participants | 61.2 [54.2 to 68.1] | 65.4 [58.6 to 72.2]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 vs Bevacizumab + FOLFIRI; Test type: Superiority or Other; Difference in Objective Response Rates = 4.3, 95% CI 2-sided [-5.5 to 14.0] — The difference was calculated as the percentage of participants with objective response in the Bevacizumab + FOLFIRI arm minus the Bevacizumab + mFOLFOX6 arm. The 95% CI was computed using normal approximation to the binomial distribution

15. Secondary Outcome: Percentage of Participants With Objective Response According to RECIST Version 1.1 in Participants With High ERCC-1 Levels
Description: Objective response was defined as CR or PR according to RECIST Version 1.1. CR was defined as disappearance of all target lesions and short-axis reduction to <10 mm of any pathological lymph nodes. PR was defined as ≥30% decrease in sum of LD of target lesions in reference to sum of LD at Baseline. Confirmation of response at a consecutive assessment was not required. The percentage of participants with CR or PR was reported. The 95% CI was computed using normal approximation to the binomial distribution.
Time Frame: From Baseline until disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 High) | Bevacizumab + FOLFIRI (ERCC-1 High)
Number analyzed (Participants) | 64 | 67
percentage of participants | 56.3 [44.1 to 68.4] | 65.7 [54.3 to 77.0]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 High) vs Bevacizumab + FOLFIRI (ERCC-1 High); Test type: Superiority or Other; Difference in Objective Response Rates = 9.4, 95% CI 2-sided [7.2 to 26.1] — [estimate comment as in outcome 14, analysis 1]

16. Secondary Outcome: Percentage of Participants With Objective Response According to RECIST Version 1.1 in Participants With Low ERCC-1 Levels
Description: as for outcome 15
Time Frame: From Baseline until disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 Low) | Bevacizumab + FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 124 | 120
percentage of participants | 63.7 [55.2 to 72.2] | 65.8 [57.3 to 74.3]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 Low) vs Bevacizumab + FOLFIRI (ERCC-1 Low); Test type: Superiority or Other; Difference in Objective Response Rates = 2.1, 95% CI 2-sided [-9.9 to 14.1] — [estimate comment as in outcome 14, analysis 1]

17. Secondary Outcome: Percentage of Participants With Objective Response According to RECIST Version 1.1 in Participants With High ERCC-1 Levels Versus Participants With Low ERCC-1 Levels
Description: as for outcome 15
Time Frame: From Baseline until disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 131 | 244
percentage of participants | 61.1 [52.7 to 69.4] | 64.8 [58.8 to 70.7]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) vs Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low); Test type: Superiority or Other; Difference in Objective Response Rates = -3.7, 95% CI 2-sided [-14.0 to 6.6] — The difference was calculated as the percentage of participants with objective response in the ERCC-1 High subgroup minus the ERCC-1 Low subgroup. The 95% CI was computed using normal approximation to the binomial distribution

18. Secondary Outcome: Percentage of Participants With Disease Control According to RECIST Version 1.1
Description: Disease control was defined as CR, PR, or stable disease (SD) according to RECIST Version 1.1. CR was defined as disappearance of all target lesions and short-axis reduction to <10 mm of any pathological lymph nodes. PR was defined as ≥30% decrease in sum of LD of target lesions in reference to sum of LD at Baseline. Confirmation of response at a consecutive assessment was not required. SD was defined as neither sufficient shrinkage to quality for PR nor sufficient increase to qualify for disease progression (≥20% increase in sum of LD of target lesions plus absolute increase ≥5 mm) in reference to the smallest sum of LD on study. The percentage of participants with CR, PR, or SD was reported. The 95% CI was computed using normal approximation to the binomial distribution.
Time Frame: From Baseline until disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 | Bevacizumab + FOLFIRI
Number analyzed (Participants) | 188 | 188
percentage of participants | 93.1 [89.5 to 96.7] | 91.0 [86.9 to 95.1]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 vs Bevacizumab + FOLFIRI; Test type: Superiority or Other; Difference in Disease Control Rates = 2.1, 95% CI 2-sided [-7.6 to 3.3] — The difference was calculated as the percentage of participants with disease control in the Bevacizumab + FOLFIRI arm minus the Bevacizumab + mFOLFOX6 arm. The 95% CI was computed using normal approximation to the binomial distribution

19. Secondary Outcome: Percentage of Participants With Disease Control According to RECIST Version 1.1 in Participants With High ERCC-1 Levels
Description: Disease control was defined as CR, PR, or SD according to RECIST Version 1.1. CR was defined as disappearance of all target lesions and short-axis reduction to <10 mm of any pathological lymph nodes. PR was defined as ≥30% decrease in sum of LD of target lesions in reference to sum of LD at Baseline. Confirmation of response at a consecutive assessment was not required. SD was defined as neither sufficient shrinkage to quality for PR nor sufficient increase to qualify for disease progression (≥20% increase in sum of LD of target lesions plus absolute increase ≥5 mm) in reference to the smallest sum of LD on study. The percentage of participants with CR, PR, or SD was reported. The 95% CI was computed using normal approximation to the binomial distribution.
Time Frame: From Baseline until disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 High) | Bevacizumab + FOLFIRI (ERCC-1 High)
Number analyzed (Participants) | 64 | 67
percentage of participants | 93.8 [87.8 to 99.7] | 85.1 [76.5 to 93.6]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 High) vs Bevacizumab + FOLFIRI (ERCC-1 High); Test type: Superiority or Other; Difference in Disease Control Rates = -8.7, 95% CI 2-sided [-19.1 to 1.7] — [estimate comment as in outcome 18, analysis 1]

20. Secondary Outcome: Percentage of Participants With Disease Control According to RECIST Version 1.1 in Participants With Low ERCC-1 Levels
Description: as for outcome 19
Time Frame: From Baseline until disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 Low) | Bevacizumab + FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 124 | 120
percentage of participants | 92.7 [88.2 to 97.3] | 95.0 [91.1 to 98.9]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 Low) vs Bevacizumab + FOLFIRI (ERCC-1 Low); Test type: Superiority or Other; Difference in Disease Control Rates = 2.3, 95% CI 2-sided [-3.7 to 8.3] — [estimate comment as in outcome 18, analysis 1]

21. Secondary Outcome: Percentage of Participants With Disease Control According to RECIST Version 1.1 in Participants With High ERCC-1 Levels Versus Participants With Low ERCC-1 Levels
Description: as for outcome 19
Time Frame: From Baseline until disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 131 | 244
percentage of participants | 89.3 [84.0 to 94.6] | 93.9 [90.8 to 96.9]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) vs Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low); Test type: Superiority or Other; Difference in Disease Control Rates = -4.5, 95% CI 2-sided [-10.6 to 1.5] — The difference was calculated as the percentage of participants with disease control in the ERCC-1 High subgroup minus the ERCC-1 Low subgroup. The 95% CI was computed using normal approximation to the binomial distribution

22. Secondary Outcome: Percentage of Participants With Liver Metastasis Resection
Description: The timing of resective surgery was not defined in the protocol and was left at the discretion of the Investigator. Resection was classified as R0, R1, or R2 following surgery. R0 was defined as complete resection with clear margins ≥1 mm. R1 was defined as the presence of exposed tumor or histologically detected tumor cells at the line of transection, or <1 mm microscopic margins. In the case of use of radiofrequency ablation or cryotherapy, the resection was considered as R1. R2 was defined as macroscopic positive margins or incomplete resection at time of surgery. The percentage of participants with resection of liver or liver plus lymph node metastases was reported. The 95% CI was computed using normal approximation to the binomial distribution.
Time Frame: At time of resective surgery during study (maximum up to 45 months overall)
Population: ITT Population; only those participants with liver or liver plus lymph node metastases were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 | Bevacizumab + FOLFIRI
Number analyzed (Participants) | 67 | 55
percentage of participants | 14.9 [6.4 to 23.5] | 10.9 [2.7 to 19.1]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 vs Bevacizumab + FOLFIRI; Test type: Superiority or Other; Difference in Resection Rates = -4.0, 95% CI 2-sided [-15.9 to 7.8] — The difference was calculated as the percentage of participants with resection in the Bevacizumab + FOLFIRI arm minus the Bevacizumab + mFOLFOX6 arm. The 95% CI was computed using normal approximation to the binomial distribution

23. Secondary Outcome: Percentage of Participants With Complete Liver Metastasis Resection
Description: The timing of resective surgery was not defined in the protocol and was left at the discretion of the Investigator. Resection was classified as R0, R1, or R2 following surgery. R0 was defined as complete resection with clear margins ≥1 mm. The percentage of participants with R0 resection of liver or liver plus lymph node metastases was reported. The 95% CI was computed using normal approximation to the binomial distribution.
Time Frame: At time of resective surgery during study (maximum up to 45 months overall)
Population: ITT Population; only those participants with liver or liver plus lymph node metastases were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 | Bevacizumab + FOLFIRI
Number analyzed (Participants) | 67 | 55
percentage of participants | 11.9 [4.2 to 19.7] | 5.5 [0.0 to 11.5]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 vs Bevacizumab + FOLFIRI; Test type: Superiority or Other; Difference in Complete Resection Rates = -6.5, 95% CI 2-sided [-16.3 to 3.3] — The difference was calculated as the percentage of participants with complete resection in the Bevacizumab + FOLFIRI arm minus the Bevacizumab + mFOLFOX6 arm. The 95% CI was computed using normal approximation to the binomial distribution

24. Secondary Outcome: Percentage of Participants With Liver Metastasis Resection in Participants With High ERCC-1 Levels
Description: as for outcome 22
Time Frame: At time of resective surgery during study (maximum up to 45 months overall)
Population: ITT Population; only those participants with liver or liver plus lymph node metastases were included in the analysis. The "Number of Participants Analyzed" reflects the number of evaluable participants for the outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 High) | Bevacizumab + FOLFIRI (ERCC-1 High)
Number analyzed (Participants) | 17 | 15
percentage of participants | 17.6 [0.0 to 35.8] | 6.7 [0.0 to 19.3]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 High) vs Bevacizumab + FOLFIRI (ERCC-1 High); Test type: Superiority or Other; Difference in Resection Rates = -11.0, 95% CI 2-sided [-33.1 to 11.1] — [estimate comment as in outcome 22, analysis 1]

25. Secondary Outcome: Percentage of Participants With Complete Liver Metastasis Resection in Participants With High ERCC-1 Levels
Description: as for outcome 23
Time Frame: At time of resective surgery during study (maximum up to 45 months overall)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 High) | Bevacizumab + FOLFIRI (ERCC-1 High)
Number analyzed (Participants) | 17 | 15
percentage of participants | 17.6 [0.0 to 35.8] | 6.7 [0.0 to 19.3]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 High) vs Bevacizumab + FOLFIRI (ERCC-1 High); Test type: Superiority or Other; Difference in Complete Resection Rates = -11.0, 95% CI 2-sided [-33.1 to 11.1] — [estimate comment as in outcome 23, analysis 1]

26. Secondary Outcome: Percentage of Participants With Liver Metastasis Resection in Participants With Low ERCC-1 Levels
Description: as for outcome 22
Time Frame: At time of resective surgery during study (maximum up to 45 months overall)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 Low) | Bevacizumab + FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 124 | 120
percentage of participants | 10.5 [5.1 to 15.9] | 7.5 [2.8 to 12.2]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 Low) vs Bevacizumab + FOLFIRI (ERCC-1 Low); Test type: Superiority or Other; Difference in Resection Rates = -3.0, 95% CI 2-sided [-10.1 to 4.2] — [estimate comment as in outcome 22, analysis 1]

27. Secondary Outcome: Percentage of Participants With Complete Liver Metastasis Resection in Participants With Low ERCC-1 Levels
Description: as for outcome 23
Time Frame: At time of resective surgery during study (maximum up to 45 months overall)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX6 (ERCC-1 Low) | Bevacizumab + FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 124 | 120
percentage of participants | 8.9 [3.9 to 13.9] | 3.3 [0.1 to 6.5]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX6 (ERCC-1 Low) vs Bevacizumab + FOLFIRI (ERCC-1 Low); Test type: Superiority or Other; Difference in Complete Resection Rates = -5.5, 95% CI 2-sided [-11.5 to 0.4] — [estimate comment as in outcome 23, analysis 1]

28. Secondary Outcome: Percentage of Participants With Liver Metastasis Resection in Participants With High ERCC-1 Levels Versus Participants With Low ERCC-1 Levels
Description: as for outcome 22
Time Frame: At time of resective surgery during study (maximum up to 45 months overall)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 131 | 244
percentage of participants | 4.6 [1.0 to 8.2] | 9.0 [5.4 to 12.6]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) vs Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low); Test type: Superiority or Other; Difference in Resection Rates = -4.4, 95% CI 2-sided [-9.5 to 0.6] — The difference was calculated as the percentage of participants with resection in the ERCC-1 High subgroup minus the ERCC-1 Low subgroup. The 95% CI was computed using normal approximation to the binomial distribution

29. Secondary Outcome: Percentage of Participants With Complete Liver Metastasis Resection in Participants With High ERCC-1 Levels Versus Participants With Low ERCC-1 Levels
Description: as for outcome 23
Time Frame: At time of resective surgery during study (maximum up to 45 months overall)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) | Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low)
Number analyzed (Participants) | 131 | 244
percentage of participants | 4.6 [1.0 to 8.2] | 6.1 [3.1 to 9.2]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 High) vs Bevacizumab + mFOLFOX/FOLFIRI (ERCC-1 Low); Test type: Superiority or Other; Difference in Complete Resection Rates = -1.6, 95% CI 2-sided [-6.2 to 3.1] — The difference was calculated as the percentage of participants with complete resection in the ERCC-1 High subgroup minus the ERCC-1 Low subgroup. The 95% CI was computed using normal approximation to the binomial distribution

30. Secondary Outcome: PFS According to RECIST Version 1.1 in Participants With Wild-Type V-Ki-ras2 Kirsten Rat Sarcoma Viral Oncogene Homolog (KRAS) Versus Participants With Mutant KRAS
Description: as for outcome 2
Time Frame: From Baseline until death or disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX/FOLFIRI (KRAS Wild-Type): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 or bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Depending on the regimen to which the participant was randomized, bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin or irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with wild-type KRAS at Baseline were included in separate analyses.
- Bevacizumab + mFOLFOX/FOLFIRI (KRAS Mutant): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 or bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Depending on the regimen to which the participant was randomized, bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin or irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with mutant KRAS at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (KRAS Wild-Type) | Bevacizumab + mFOLFOX/FOLFIRI (KRAS Mutant)
Number analyzed (Participants) | 208 | 128
months | 12.45 [10.48 to 14.06] | 10.94 [8.77 to 12.35]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (KRAS Wild-Type) vs Bevacizumab + mFOLFOX/FOLFIRI (KRAS Mutant); Analysis stratified by high/low ERCC-1 level and region of enrollment; Test type: Superiority or Other; p = 0.0593, Log Rank — P-value (relative to KRAS Wild-Type subgroup) based on two-sided stratified log rank test and not adjusted for multiple comparisons; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.99 to 1.69] — HR (relative to KRAS Wild-Type subgroup) was estimated by Cox regression

31. Secondary Outcome: OS in Participants With High VEGF-A Levels Versus Participants With Low VEGF-A Levels
Description: as for outcome 10
Time Frame: From Baseline until death (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High): Participants with untreated mCRC who were candidates for first-line therapy received bevacizumab plus mFOLFOX6 or bevacizumab plus FOLFIRI until disease progression or unacceptable toxicity. Depending on the regimen to which the participant was randomized, bevacizumab was given as 5 mg/kg, leucovorin as 400 mg/m^2, oxaliplatin as 85 mg/m^2, irinotecan as 180 mg/m^2, and 5-fluorouracil as 400 mg/m^2 bolus followed by 2400 mg/m^2 continuous 46-hour infusion. All treatments were administered via IV infusion and started on Day 1 of each 2-week cycle. Participants could be transitioned to oral capecitabine in the event of unacceptable toxicity to oxaliplatin or irinotecan and given as 850 or 1000 mg/m^2 twice a day on Days 1 to 14, with bevacizumab continued in 3-week cycles. Participants with VEGF-A level >5 pg/mL at Baseline were included in separate analyses.
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low)
Number analyzed (Participants) | 185 | 185
months | 22.83 [18.76 to 27.27] | 27.93 [24.97 to 36.01]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) vs Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low); Analysis stratified by high/low ERCC-1 level and region of enrollment; Test type: Superiority or Other; p = 0.0020, Log Rank — [p-value comment as in outcome 5, analysis 1]; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [1.20 to 2.24] — HR (relative to VEGF-A Low subgroup) was estimated by Cox regression

32. Secondary Outcome: OS in Participants With Wild-Type KRAS Versus Participants With Mutant KRAS
Description: as for outcome 10
Time Frame: From Baseline until death (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (KRAS Wild-Type) | Bevacizumab + mFOLFOX/FOLFIRI (KRAS Mutant)
Number analyzed (Participants) | 208 | 128
months | 28.75 [24.77 to 36.73] | 24.64 [19.98 to 26.94]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (KRAS Wild-Type) vs Bevacizumab + mFOLFOX/FOLFIRI (KRAS Mutant); Analysis stratified by high/low ERCC-1 level and region of enrollment; Test type: Superiority or Other; p = 0.0955, Log Rank — [p-value comment as in outcome 30, analysis 1]; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.95 to 1.88] — HR (relative to KRAS Wild-Type subgroup) was estimated by Cox regression

33. Secondary Outcome: Percentage of Participants With Objective Response According to RECIST Version 1.1 in Participants With High VEGF-A Levels Versus Participants With Low VEGF-A Levels
Description: as for outcome 15
Time Frame: From Baseline until disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low)
Number analyzed (Participants) | 185 | 185
percentage of participants | 60.5 [53.5 to 67.6] | 66.5 [59.7 to 73.3]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) vs Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low); Test type: Superiority or Other; Difference in Objective Response Rates = -5.9, 95% CI 2-sided [-15.7 to 3.8] — The difference was calculated as the percentage of participants with objective response in the VEGF-A High subgroup minus the VEGF-A Low subgroup. The 95% CI was computed using normal approximation to the binomial distribution

34. Secondary Outcome: Percentage of Participants With Objective Response According to RECIST Version 1.1 in Participants With Wild-Type KRAS Versus Participants With Mutant KRAS
Description: as for outcome 15
Time Frame: From Baseline until disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (KRAS Wild-Type) | Bevacizumab + mFOLFOX/FOLFIRI (KRAS Mutant)
Number analyzed (Participants) | 208 | 128
percentage of participants | 66.3 [59.9 to 72.8] | 60.9 [52.5 to 69.4]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (KRAS Wild-Type) vs Bevacizumab + mFOLFOX/FOLFIRI (KRAS Mutant); Test type: Superiority or Other; Difference in Objective Response Rates = -5.4, 95% CI 2-sided [-16.0 to 5.2] — The difference was calculated as the percentage of participants with objective response in the KRAS Mutant subgroup minus the KRAS Wild-Type subgroup. The 95% CI was computed using normal approximation to the binomial distribution

35. Secondary Outcome: Percentage of Participants With Disease Control According to RECIST Version 1.1 in Participants With High VEGF-A Levels Versus Participants With Low VEGF-A Levels
Description: as for outcome 19
Time Frame: From Baseline until disease progression; assessed every 6 weeks (maximum up to 45 months overall)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low)
Number analyzed (Participants) | 185 | 185
percentage of participants | 91.9 [88.0 to 95.8] | 93.0 [89.3 to 96.7]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) vs Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low); Test type: Superiority or Other; Difference in Disease Control Rates = -1.1, 95% CI 2-sided [-6.5 to 4.3] — The difference was calculated as the percentage of participants with disease control in the VEGF-A High subgroup minus the VEGF-A Low subgroup. The 95% CI was computed using normal approximation to the binomial distribution

36. Secondary Outcome: Percentage of Participants With Liver Metastasis Resection in Participants With High VEGF-A Levels Versus Participants With Low VEGF-A Levels
Description: as for outcome 22
Time Frame: At time of resective surgery during study (maximum up to 45 months overall)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low)
Number analyzed (Participants) | 185 | 185
percentage of participants | 5.9 [2.5 to 9.4] | 9.2 [5.0 to 13.4]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) vs Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low); Test type: Superiority or Other; Difference in Resection Rates = -3.2, 95% CI 2-sided [-8.6 to 2.1] — The difference was calculated as the percentage of participants with resection in the VEGF-A High subgroup minus the VEGF-A Low subgroup. The 95% CI was computed using normal approximation to the binomial distribution

37. Secondary Outcome: Percentage of Participants With Complete Liver Metastasis Resection in Participants With High VEGF-A Levels Versus Participants With Low VEGF-A Levels
Description: as for outcome 23
Time Frame: At time of resective surgery during study (maximum up to 45 months overall)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) | Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low)
Number analyzed (Participants) | 185 | 185
percentage of participants | 3.2 [0.7 to 5.8] | 8.1 [4.2 to 12.0]
Statistical Analysis 1: Comparison: Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A High) vs Bevacizumab + mFOLFOX/FOLFIRI (VEGF-A Low); Test type: Superiority or Other; Difference in Complete Resection Rates = -4.9, 95% CI 2-sided [-9.6 to -0.2] — The difference was calculated as the percentage of participants with complete resection in the VEGF-A High subgroup minus the VEGF-A Low subgroup. The 95% CI was computed using normal approximation to the binomial distribution

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (AEs): Baseline until 3 months after last dose or study discontinuation/termination (up to 45 months overall); Other AEs: Baseline until 28 days after last dose or study discontinuation/termination (up to 45 months overall).
Description: Safety Population: All randomized participants who received at least one partial or complete dose of study drug.
Arm/Group | Bevacizumab + mFOLFOX6 | Bevacizumab + FOLFIRI
Serious Adverse Events (participants affected / at risk) | 79/185 | 87/183
Other Adverse Events (participants affected / at risk) | 185/185 | 181/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + mFOLFOX6 (N=185) | Bevacizumab + FOLFIRI (N=183)
Diarrhoea (Gastrointestinal disorders) | 6 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 6
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 7
Intestinal obstruction (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Oesophageal motility disorder (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Anal fistula (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 4 | 3
Pneumonia (Infections and infestations) | 3 | 7
Cellulitis (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Candida sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Perineal abscess (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 8 | 5
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1
Chest pain (General disorders) | 3 | 4
Pyrexia (General disorders) | 3 | 4
Device dislocation (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Device malfunction (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 3
Gait disturbance (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Hypotension (Vascular disorders) | 5 | 1
Hypertension (Vascular disorders) | 3 | 6
Arterial thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 4
Embolism venous (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 3
Atrial thrombosis (Cardiac disorders) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Aphonia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Biloma (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Platelet count decreased (Investigations) | 2 | 0
Weight decreased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Proteinuria (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colostomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + mFOLFOX6 (N=185) | Bevacizumab + FOLFIRI (N=183)
Diarrhoea (Gastrointestinal disorders) | 99 | 123
Nausea (Gastrointestinal disorders) | 106 | 109
Constipation (Gastrointestinal disorders) | 63 | 65
Vomiting (Gastrointestinal disorders) | 58 | 57
Abdominal pain (Gastrointestinal disorders) | 39 | 54
Stomatitis (Gastrointestinal disorders) | 35 | 38
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 17 | 18
Dyspepsia (Gastrointestinal disorders) | 19 | 14
Rectal haemorrhage (Gastrointestinal disorders) | 11 | 18
Abdominal pain upper (Gastrointestinal disorders) | 8 | 15
Oral pain (Gastrointestinal disorders) | 8 | 14
Haemorrhoids (Gastrointestinal disorders) | 6 | 16
Proctalgia (Gastrointestinal disorders) | 7 | 13
Dry mouth (Gastrointestinal disorders) | 7 | 11
Abdominal distension (Gastrointestinal disorders) | 5 | 12
Dysphagia (Gastrointestinal disorders) | 10 | 2
Fatigue (General disorders) | 105 | 104
Mucosal inflammation (General disorders) | 37 | 51
Pyrexia (General disorders) | 18 | 29
Asthenia (General disorders) | 21 | 18
Oedema peripheral (General disorders) | 18 | 18
Temperature intolerance (General disorders) | 34 | 1
Chest pain (General disorders) | 15 | 10
Chills (General disorders) | 10 | 10
Influenza like illness (General disorders) | 10 | 6
Neuropathy peripheral (Nervous system disorders) | 85 | 23
Headache (Nervous system disorders) | 31 | 38
Dysgeusia (Nervous system disorders) | 33 | 31
Paraesthesia (Nervous system disorders) | 35 | 15
Peripheral sensory neuropathy (Nervous system disorders) | 35 | 12
Dizziness (Nervous system disorders) | 15 | 28
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 41 | 59
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 26
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 | 21
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 14 | 18
Hiccups (Respiratory, thoracic and mediastinal disorders) | 8 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Decreased appetite (Metabolism and nutrition disorders) | 56 | 55
Hypokalaemia (Metabolism and nutrition disorders) | 36 | 33
Dehydration (Metabolism and nutrition disorders) | 28 | 27
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 23
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 61
Dry skin (Skin and subcutaneous tissue disorders) | 27 | 26
Rash (Skin and subcutaneous tissue disorders) | 19 | 26
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 24 | 18
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 18 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 10
Neutropenia (Blood and lymphatic system disorders) | 65 | 86
Anaemia (Blood and lymphatic system disorders) | 25 | 34
Thrombocytopenia (Blood and lymphatic system disorders) | 44 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 25
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 19
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 11
Weight decreased (Investigations) | 33 | 29
Neutrophil count decreased (Investigations) | 33 | 23
Platelet count decreased (Investigations) | 24 | 3
White blood cell count decreased (Investigations) | 15 | 9
Insomnia (Psychiatric disorders) | 29 | 35
Depression (Psychiatric disorders) | 24 | 18
Anxiety (Psychiatric disorders) | 19 | 20
Hypertension (Vascular disorders) | 61 | 54
Urinary tract infection (Infections and infestations) | 18 | 20
Upper respiratory tract infection (Infections and infestations) | 15 | 18
Sinusitis (Infections and infestations) | 9 | 13
Proteinuria (Renal and urinary disorders) | 38 | 39
Vision blurred (Eye disorders) | 13 | 12
Lacrimation increased (Eye disorders) | 4 | 10
Infusion related reaction (Injury, poisoning and procedural complications) | 15 | 8
Hypersensitivity (Immune system disorders) | 10 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.